CLINICAL TRIAL: NCT06695195
Title: A Randomized Controlled Trial of Oral CBD for the Treatment of Upper Extremity Musculoskeletal Pain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brent DeGeorge (Other)
Collaborators: The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor-Investigator, Brent DeGeorge, Associate Professor of Plastic Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301881
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-12

CONDITIONS: Upper Extremity Muscle Pain; Upper Extremity Bone Pain; Upper Extremity Pain
Keywords: Wrist Muscular Pain; Forearm Bone Pain; Forearm Muscular Pain; Hand Pain; CBD; oral CBD; Upper Arm Muscular Pain; Upper Arm Bone Pain; Wrist Joint Pain; Wrist Bone Pain; Forearm Joint Pain; Upper Arm Joint Pain
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: The study design will be a double-blind, randomized controlled trial with crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral CBD (Experimental): Oral CBD 25 mg capsules taken twice each day for 4 weeks.
  Interventions: Drug: Cannabidiol (CBD)
- Placebo (Placebo Comparator): Oral placebo capsules taken twice each day for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) — 25 mg capsule twice daily
  Other Names: Green Valley Nutrition, LLC; Cannabidiol
  Arms: Oral CBD
Drug: Placebo — 25 mg capsule twice daily
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the use of cannabidiol (CBD) capsules as a treatment for musculoskeletal pain. CBD is commonly being used as an over-the-counter treatment for musculoskeletal pain. Clinical trials have demonstrated a pain-relief benefit for hand and wrist osteoarthritis with topical CBD, however patients prefer oral CBD and no clinical trial has been performed to establish efficacy of oral CBD in humans for upper extremity musculoskeletal pain. The main questions it aims to answer are:

Is CBD more effective than placebo at relieving pain for upper extremity musculoskeletal pain ? Is CBD safe for participants with upper extremity musculoskeletal pain?

Participants will:

take 4 weeks of daily CBD capsules take 4 weeks of daily placebo capsules answer surveys about how they are feeling and functioning.

Participants will [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

DETAILED DESCRIPTION:
This randomized controlled trial of CBD will investigate the therapeutic potential of CBD as an oral treatment for the treatment of pain of upper extremity musculoskeletal pain. Rationale: CBD is commonly being used as an over-the-counter treatment for musculoskeletal pain. Clinical trials have demonstrated a pain-relief benefit for hand and wrist osteoarthritis with topical CBD, however patients prefer oral CBD and no clinical trial has been performed to establish efficacy of oral CBD in humans for upper extremity musculoskeletal pain. Hypothesis: CBD is more effective than placebo for relieving pain and improving patient-reported outcomes for upper extremity musculoskeletal pain.

Study Design: The study design will be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 4 weeks of the CBD or control and then crossover to the other condition for 4 additional weeks. Patients will take one oral capsule twice daily, once in the morning and once in the evening. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 years or older.
4. Daily visual analog pain score >5/10 and <9/10.
5. Duration of pain for greater than or equal to 3 months.
6. Presence of physician-diagnosed musculoskeletal pain in the upper extremities, including bone or joint-related pain, tendon or ligament-related pain, muscle-related pain, or fibromyalgia or physician-diagnosed postoperative pain in a discrete body region, limited to upper extremities.
7. For females, must be willing to use an approved form of birth control during this study. Acceptable forms of birth control:

   * Norplant
   * Sterilization
   * IUD (intrauterine device)
   * Birth Control Patch
   * Depo-Provera

   The following may be used if combined with other birth control methods:
   * Condoms
   * Diaphragm
   * Jellies or foam
   * Sponge
   * Cervical cap
8. For males, must be willing to not father a baby for the duration of the study and for 90 days after the last dose of study drug, or donate to a sperm bank during this time. Must be willing to use an approved form of birth control during this time. Acceptable forms of birth control:

   * Condoms
   * Sterilization

Exclusion Criteria:

1. Subject does not speak or read English fluently.
2. Subject is blind.
3. Severe cardiac, pulmonary, liver and /or renal disease, or any other major organ dysfunction.
4. Subject with a history of symptoms (e.g., dizziness, light-headedness, blurred vision, palpitations, weakness, syncope) related to a drop in blood pressure due to postural changes.
5. Coumadin use at time of screening.
6. History of mental illness.
7. Subjects who are incarcerated.
8. Subjects who satisfy any DSM-V criteria for current psychiatric illness such as bipolar disorder, depression, anxiety, schizophrenia, psychosis, substance use disorder or any other psychiatric diagnosis
9. Subjects who have used intra-articular corticosteroids 30 days prior to screening.
10. History of drug or substance abuse.
11. Pre-existing CBD product usage currently (or within the prior 3 months) using recreational or medicinal cannabis, any cannabinoid-based medications, and is unwilling to abstain for the duration of the study.
12. Subject has had a corticosteroid injection ≤ 60 days prior.
13. Subjects who are unwilling to agree to no opioid medications or topical analgesic medications during the study period.
14. Any woman of child bearing potential or male patient's partner unwilling to ensure that they or their partner use effective contraception, for example, hormonal contraception, double barrier, intra-uterine device, during the study and for females, through 30 days thereafter, and for males, three months thereafter.
15. Any male not willing to avoid donating sperm during the duration of the study treatment period and for three months thereafter.
16. Any patient with aberrant liver function as defined by either of the following:

    * ALT >5x ULN or total bilirubin>2×ULN
    * ALT or AST>3 × ULN and total bilirubin>2xULN or INR >1.5
17. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP3A4 :

    * Itraconazole,
    * Ketoconazole,
    * Azamulin,
    * Troleandomycin,
    * Verapamil,
    * John's wart,
    * Phenobarbital,
18. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP2C19:

    * Nootkatone,
    * Ticlopidine,
    * Rifampin,
    * Omeprazole),
19. Subjects taking prescription or non-prescription medication which are substrates of CYP2C8:

    * Montelukast,
    * Quercetin,
    * Phenelzine,
    * Rifampin,
    * Clopidogrel) ,
20. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates ofCYP2C9:

    * Sulfaphenazole,
    * Tienilic acid,
    * Carbamazepine,
    * Apalutamide,
    * Fluconazole,
    * Celecoxib
21. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP1A2:

    * alpha-Naphthoflavone,
    * Furafylline,
    * Phenytoin,
    * Rifampin,
    * Ritonavir,
    * smoking,
    * Teriflunomide,
    * Ciproflaoxacin,
    * oral contraceptives,
    * Allopurinol
22. Participants within 14 days of the study procedure taking prescription or non-prescription medication which are substrates of CYP2B6:

    * Sertraline,
    * Phencyclidine,
    * Thiotepa,
    * Ticlopidine,
    * Carbamazepine,
    * Efavirenez,
    * Rifampin,
    * Bupropion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain on the Visual Analog Pain (VAS) Score | Baseline and Week 4, Week 6
  The Visual Analog Pain (VAS) Score is a validated, self-reported subjective measure for measuring acute and chronic pain. Possible scores range from 0 (no pain) to 10 (worst possible pain). Change = (Week (4 or 6) Score - Baseline Score).a validated, self-report
Change from Baseline in Pain on the Visual Analog Pain (VAS) Score - Crossover Condition | Baseline and Week 4, Week 6
  The Visual Analog Pain (VAS) Score is a validated, self-reported subjective measure for measuring acute and chronic pain. Possible scores range from 0 (no pain) to 10 (worst possible pain). Change = (Week (4 or 6) Score - Baseline Score).a validated, self-report
Change from Baseline in Normal Function on the Single Assessment Numerical Evaluation (SANE) Score | Baseline and Week 4, Week 6
  The SANE Score is a self-reported subjective measure for measuring percentage of normal function. Possible scores range from 0 (most abnormal) to 100 (normal). Change = (Week (4 or 6) Score - Baseline Score)
Change from Baseline in Normal Function on the Single Assessment Numerical Evaluation (SANE) Score - Crossover Condition | Baseline and Week 4, Week 6
  The SANE Score is a self-reported subjective measure for measuring percentage of normal function. Possible scores range from 0 (most abnormal) to 100 (normal). Change = (Week (4 or 6) Score - Baseline Score)
Change from Baseline in Quality of Life on the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health-10 Score | Baseline and Week 4, Week 6
  The PROMIS Global Health-10 is a validated, self-reported subjective measure for measuring generic health related quality of life. Possible scores range from 0 (most severe impairment) to 20 (best health). Change = (Week (4 or 6) Score - Baseline Score)
Change from Baseline in Quality of Life on the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health-10 Score - Crossover Condition | Baseline and Week 4, Week 6
  The PROMIS Global Health-10 is a validated, self-reported subjective measure for measuring generic health related quality of life. Possible scores range from 0 (most severe impairment) to 20 (best health). Change = (Week (4 or 6) Score - Baseline Score)
Change from Baseline in Pain interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score | Baseline and Week 4, Week 6
  The PROMIS Pain Interference is a validated, self-reported subjective measure for measuring generic health related quality of life. Possible scores range from 0 (does not interfere) to 10 (completely interferes). Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Pain interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score - Crossover Condition | Baseline and Week 4, Week 6
  The PROMIS Pain Interference is a validated, self-reported subjective measure for measuring generic health related quality of life. Possible scores range from 0 (does not interfere) to 10 (completely interferes). Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Pain interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Upper Extremity (UE) Score | Baseline and Week 4, Week 6
  The PROMIS UE computer adaptive test is a validated computer adaptive test to assess upper extremity functional status. Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Pain interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Upper Extremity (UE) Score - Crossover Condition | Baseline and Week 4, Week 6
  The PROMIS UE computer adaptive test is a validated computer adaptive test to assess upper extremity functional status. Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Pain on the Australian/Canadian Hand Osteoarthritis (AUSCAN) Index | Baseline and Week 4, Week 6
  The AUSCAN Index is a 15-item scale measuring pain (5 items), stiffness (1 item) and function (9 items) during the preceding 48 hours. Possible scores range from 0 (none) to 4 (extreme). Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Pain on the Australian/Canadian Hand Osteoarthritis (AUSCAN) Index - Crossover Condition | Baseline and Week 4, Week 6
  The AUSCAN Index is a 15-item scale measuring pain (5 items), stiffness (1 item) and function (9 items) during the preceding 48 hours. Possible scores range from 0 (none) to 4 (extreme). Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in Disability on The Quick Disability of the Arm, Shoulder (QuickDASH) | Baseline and Week 4
  The QuickDASH is a validated, self-reported 11-item scale measuring disability. Possible scores range from 0 (no disability) to 100 (most severe disability. Change = (Week 4 Score - Baseline Score)
Change from Baseline in Disability on The Quick Disability of the Arm, Shoulder (QuickDASH) - Crossover Condition | Baseline and Week 4
  The QuickDASH is a validated, self-reported 11-item scale measuring disability. Possible scores range from 0 (no disability) to 100 (most severe disability. Change = (Week 4 Score - Baseline Score)
Change from Baseline in perseverance on the Brief Resilience Index (BRI) | Baseline and Week 4, Week 6
  The BRI is a validated, self-reported 6-item validated tool to assess for resilience. Possible scores range from 1 (low resilience) to 5 (high resilience). Change = (Week (4, 6) Score - Baseline Score)
Change from Baseline in perseverance on the Brief Resilience Index (BRI) - Crossover Condition | Baseline and Week 4, Week 6
  The BRI is a validated, self-reported 6-item validated tool to assess for resilience. Possible scores range from 1 (low resilience) to 5 (high resilience). Change = (Week (4, 6) Score - Baseline Score)

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | Through study completion, an average of 12 weeks
  Treatment-related adverse events will be reported throughout the study by self-report and clinician-driven questions at each visit
Change from Baseline in the Mean Seated Trough Cuff Systolic Blood Pressure | Baseline and Week 4
  Blood pressure (SBP and DBP) in mmHg using Sphygmomanometer will be assessed by the researchers at baseline and follow-up
Change from Baseline in Heart Rate | Baseline and Week 4
  Heartbeats per minute (BPM) will be assessed by the researchers at baseline and follow-up
Change from Baseline in the Mean Seated Trough Cuff Systolic Blood Pressure | Week 4 and Week 6
  Blood pressure (SBP and DBP) in mmHg using Sphygmomanometer will be assessed by the researchers at baseline and follow-up
Change from Baseline in Heart Rate | Week 4 and Week 6
  Heartbeats per minute (BPM) will be assessed by the researchers at baseline and follow-up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: glucose, blood urea nitrogen (BUN), Creatinine, Calcium | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: glucose, BUN, Creatinine, Calcium (mg/dL) at baseline and follow up
Change from baseline in serum liver panel parameters: Alanine transaminase (ALT), Alkaline phosphatase (ALP) and Aspartate aminotransferase (AST) | Through study completion, an average of 12 weeks
  Change from baseline in serum liver panel parameters: ALT, ALP and AST (International units per liter) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Chloride | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Chloride (umol/L) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Sodium, Potassium, Chloride, Carbon Dioxide | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Sodium, Potassium, Chloride, Carbon Dioxide (meq/L) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Bilirubin | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Bilirubin (umol/L) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Prothrombin time- International normalized ratio (PT-INR) | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Prothrombin time- International normalized ratio (PT (seconds)-INR) at baseline and follow up
Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Protein, Albumin | Through study completion, an average of 12 weeks
  Change from baseline in serum comprehensive metabolic panel (CMP) parameters: Protein, Albumin (g/dL) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: Red Blood Cells (CBC), White Blood Cells (WBC), Platelets | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: RBC, WBC, Platelets (uL) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: Hemoglobin | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: Hemoglobin (g.dL) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: Hematocrit | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: Hematocrit (percentage) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: Mean Corpuscular Volume (MCV) | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: Mean Corpuscular Volume (MCV) (pg) at baseline and follow up
Change from baseline in serum complete blood count (CBC) parameters: the amount of hemoglobin per red blood cell.(MCH) | Through study completion, an average of 12 weeks
  Change from baseline in serum complete blood count (CBC) parameters: the amount of hemoglobin per red blood cell.(MCH) (pg) at baseline and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Brent DeGeorge, MD, PhD, Principal Investigator — University of Virginia Department of Plastic Surgery
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russo E.B., Mathre M.L., Byrne A., Velin R., Bach P.J., Sanchez-Ramos J., et. al.: Chronic cannabis use in the compassionate investigational new drug program: an examination of benefits and adverse effects of legal clinical cannabis. J Cannabis Ther 2002; 2: pp. 3-57.
- [Background] Stockings E, Zagic D, Campbell G, Weier M, Hall WD, Nielsen S, Herkes GK, Farrell M, Degenhardt L. Evidence for cannabis and cannabinoids for epilepsy: a systematic review of controlled and observational evidence. J Neurol Neurosurg Psychiatry. 2018 Jul;89(7):741-753. doi: 10.1136/jnnp-2017-317168. Epub 2018 Mar 6. PMID 29511052
- [Background] Bruni N, Della Pepa C, Oliaro-Bosso S, Pessione E, Gastaldi D, Dosio F. Cannabinoid Delivery Systems for Pain and Inflammation Treatment. Molecules. 2018 Sep 27;23(10):2478. doi: 10.3390/molecules23102478. PMID 30262735
- [Background] Fader L, Scharf Z, DeGeorge BR Jr. Assessment of Medical Cannabis in Patients With Osteoarthritis of the Thumb Basal Joint. J Hand Surg Am. 2023 Mar;48(3):257-262.e1. doi: 10.1016/j.jhsa.2021.10.018. Epub 2021 Dec 8. PMID 34893392
- [Background] Ware MA, Wang T, Shapiro S, Collet JP; COMPASS study team. Cannabis for the Management of Pain: Assessment of Safety Study (COMPASS). J Pain. 2015 Dec;16(12):1233-1242. doi: 10.1016/j.jpain.2015.07.014. Epub 2015 Sep 16. PMID 26385201
- [Background] Heineman JT, Forster GL, Stephens KL, Cottler PS, Timko MP, DeGeorge BR Jr. A Randomized Controlled Trial of Topical Cannabidiol for the Treatment of Thumb Basal Joint Arthritis. J Hand Surg Am. 2022 Jul;47(7):611-620. doi: 10.1016/j.jhsa.2022.03.002. Epub 2022 May 28. PMID 35637038
- [Background] MacCallum CA, Russo EB. Practical considerations in medical cannabis administration and dosing. Eur J Intern Med. 2018 Mar;49:12-19. doi: 10.1016/j.ejim.2018.01.004. Epub 2018 Jan 4. PMID 29307505
- [Background] Arzimanoglou A, Brandl U, Cross JH, Gil-Nagel A, Lagae L, Landmark CJ, Specchio N, Nabbout R, Thiele EA, Gubbay O, The Cannabinoids International Experts Panel; Collaborators. Epilepsy and cannabidiol: a guide to treatment. Epileptic Disord. 2020 Feb 1;22(1):1-14. doi: 10.1684/epd.2020.1141. PMID 32096470
- [Background] Chen JW, Borgelt LM, Blackmer AB. Cannabidiol: A New Hope for Patients With Dravet or Lennox-Gastaut Syndromes. Ann Pharmacother. 2019 Jun;53(6):603-611. doi: 10.1177/1060028018822124. Epub 2019 Jan 8. PMID 30616356
- [Background] Mechoulam R, Hanus L. Cannabidiol: an overview of some chemical and pharmacological aspects. Part I: chemical aspects. Chem Phys Lipids. 2002 Dec 31;121(1-2):35-43. doi: 10.1016/s0009-3084(02)00144-5. PMID 12505688
- [Background] Baron EP, Lucas P, Eades J, Hogue O. Patterns of medicinal cannabis use, strain analysis, and substitution effect among patients with migraine, headache, arthritis, and chronic pain in a medicinal cannabis cohort. J Headache Pain. 2018 May 24;19(1):37. doi: 10.1186/s10194-018-0862-2. PMID 29797104
- [Background] Brat GA, Agniel D, Beam A, Yorkgitis B, Bicket M, Homer M, Fox KP, Knecht DB, McMahill-Walraven CN, Palmer N, Kohane I. Postsurgical prescriptions for opioid naive patients and association with overdose and misuse: retrospective cohort study. BMJ. 2018 Jan 17;360:j5790. doi: 10.1136/bmj.j5790. PMID 29343479
- [Background] Wolf JM, Atroshi I, Zhou C, Karlsson J, Englund M. Sick Leave After Surgery for Thumb Carpometacarpal Osteoarthritis: A Population-Based Study. J Hand Surg Am. 2018 May;43(5):439-447. doi: 10.1016/j.jhsa.2017.11.019. Epub 2018 Feb 7. PMID 29428245